CLINICAL TRIAL: NCT05158309
Title: Aalborg University, Aalborg, Denmark
Brief Title: Measuring and Modulating Changes in EEG Resting State Functional Connectivity During Short-term and Long-term Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Collaborators: Danish National Research Foundation (Other); European Commission (Other)
Responsible Party: Principal Investigator, Najah Al Hajri, Principal investigator, Aalborg University
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: N-20190057
Record Dates: First submitted 2021-12-13; First posted 2021-12-15 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Prolonged Pain, EEG, Resting State Functional Connectivity

STUDY DESIGN:
Intervention Model Description: Participants experienced both experimental (capsaicin) condition and placebo conditions. Due to the long-lasting effects of capsaicin after 24 hours of application, placebo condition always preceded the capsaicin condition.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Capsaicin (Experimental): Capsaicin condition: in this condition participants received pain using a (5x10 cm) 8% topical capsaicin patch on the volar part of the dominant right forearm.
  Interventions: Other: 8% Capsaicin patch
- Placebo (Placebo Comparator): Placebo condition: participants received no pain.
  Interventions: Other: placebo patch

INTERVENTIONS:
Other: 8% Capsaicin patch — Cutaneous pain was induced using a (5x10 cm) 8% topical capsaicin patch (transdermal patch, 'Qutenza', Astellas) on the volar part of the dominant right forearm (5 cm from the wrist) of each participant.
  Arms: Capsaicin
Other: placebo patch — A transparent patch with no formulation or effect but the same size of the capsaicin patch was applied to the same location.
  Arms: Placebo

SUMMARY:
Background and aims: Experimental prolonged pain models can shed more light on the cortical mechanisms involved in the transition from acute to chronic pain including changes in resting state functional connectivity (rsFC). This experiment aimed at examining the effect of 24-hour-capsaicin application on the rsFC of the default mode network (DMN), a prominent network in the dynamic pain connectome.

Methods: Electroencephalographic (EEG) rsFC measured by Granger causality was acquired at baseline, 1-hour, and 24-hour following the initial patch application (placebo or capsaicin). After 24 hours, the patch was cooled down then heated up to assess rsFC changes in response to pain relief and facilitation. Pain was induced using a topical capsaicin patch (or placebo as control) on the right forearm and assessed on a 0-10 numerical rating scale (NRS).

ELIGIBILITY:
Inclusion Criteria:

Healthy men and women, age 19-44, right-handed (assessed using the Edinburgh Handedness Inventory, speak and understand English.

Exclusion Criteria:

1. Chili allergies
2. History of chronic pain or current acute pain
3. Present or previous neurologic such as epilepsy, Alzheimer disease, dementia, stroke, migraine and other headache disorders, multiple sclerosis, Parkinson's disease, neuroinfections, brain tumours and head trauma.
4. Present or previous musculoskeletal disorders such muscle/tendon strain, ligament sprain tension,tendonitis, degenerative disc disease, mechanical back syndrome, and ruptured/herniated disc.
5. Present or previous mental illnesses such as depression, bipolar disorder, and schizophrenia.
6. Pregnancy
7. Current use of medications that may affect the trial (e.g. pain relieving medication and anti-inflammatory medication)
8. Using hair products that may interfere with EEG conductance such as gel, except for shampoo, prior to the trial.
9. Drug addiction defined as the use of cannabis, opioids or other drugs
10. Consumption of alcohol, caffeine, or tobacco 6 hours before the experimental onset
11. Lack of ability to cooperate -

Ages: 19 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2021-05-31 (Actual); Primary Completion 2021-11-06 (Actual); Study Completion 2021-11-06 (Actual)

PRIMARY OUTCOMES:
Change in resting state functional connectivity | Granger causality is assessed at 5 time points for each condition (capsaicin or placebo): baseline, 1 hour, 24 hours, 24 hours, cooling at 24hours, and heating at 24 hours.
  resting state functional connectivity is assessed using Granger causality. It can take on any value starting with "0" representing no connectivity. Higher granger causality scores indicate higher connectivity.
Change in Subjective pain intensity | Intensity is assessed at 5 time points for each condition (capsaicin or placebo): baseline, 1 hour, 24 hours, cooling at 24hours, and heating at 24 hours.
  Intensity rated by the participants on a numerical rating scale anchoring from 0 "no pain" to 10 "the worst imaginable pain" . Higher numerical rating scores indicate higher pain intensity.

SECONDARY OUTCOMES:
Change in Pain sensitivity (Warmth detection threshold) | Warmth detection threshold is assessed at 3 time points for each condition (capsaicin or placebo): baseline, 1 hour, and 24 hours.
  Warmth detection threshold is assessed using a thermal stimulator probe (3 × 3 cm, Pathway Medoc Ltd, Israel). Higher threshold scores indicate less sensitivity.
  .
Change in Pain sensitivity ( Cold detection threshold). | Warmth detection threshold is assessed at 3 time points for each condition (capsaicin or placebo): baseline, 1 hour, and 24 hours.
  Cold detection threshold is assessed using a thermal stimulator probe (3 × 3 cm, Pathway Medoc Ltd, Israel). Higher threshold scores indicate less sensitivity.
Change in Pain sensitivity ( Heat pain threshold). | Heat pain threshold is assessed at 3 time points for each condition (capsaicin or placebo): baseline, 1 hour, and 24 hours.
  Heat detection threshold is assessed using a thermal stimulator probe (3 × 3 cm, Pathway Medoc Ltd, Israel). Higher threshold scores indicate less sensitivity.
Change in Pain sensitivity ( Cold pain thresholds). | Cold pain threshold is assessed at 3 time points for each condition (capsaicin or placebo): baseline, 1 hour, and 24 hours.
  Cold pain threshold is assessed using a thermal stimulator probe (3 × 3 cm, Pathway Medoc Ltd, Israel). Higher threshold scores indicate less sensitivity.
Change in Pain sensitivity ( Mechanical pain thresholds). | Mechanical pain threshold is assessed at 3 time points for each condition (capsaicin or placebo): baseline, 1 hour, and 24 hours.
  Mechanical pain thresholds was assessed using a set of seven weighted pinprick stimulators consisting of steel tubes ending with a tip contact area of 0.25 mm diameter and excreting forces of 0.8, 1.6, 3.2, 6.4, 12.8, 25.6, and 51.2 g. Higher threshold scores indicate less sensitivity.
Pain vigilance | It is assessed at baseline and after 24 hours for each condition (capsaicin or placebo).
  Pain Vigilance and Awareness Questionnaire (PVAQ). This questionnaire consists of 16 items evaluating preoccupation and attention to one's pain over the past two weeks, rated between 0 = "never" and 5 = "always", with a maximum score of 80. The higher the scores, the higher the preoccupation with pain.
Pain Catastrophizing | It is assessed at baseline and after 24 hours for each condition (capsaicin or placebo).
  Scale (PCS). This questionnaire comprises 13 items assessed on a 5-point scale ranging from 0 = "not at all" to 4 = "all the time", with a maximum score of 52. It evaluates three scales of catastrophizing: rumination, magnification, and helplessness. Ratings reflect the degree to which specific thoughts and feelings are present when experiencing pain over the last three months. Higher scores indicate a higher degree of pain catastrophizing.
Sleep quality assessment | It is assessed at baseline and after 24 hours for each condition (capsaicin or placebo).
  Pittsburgh Sleep Quality Index (PSQI). This questionnaire determines sleep quality and sleep patterns across seven areas: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction over the last month. These areas are evaluated on a scale ranging from 0 = "no difficulty" to 3 = "severe difficulty," with a maximum score of 21. Higher scores reflect poor sleep quality.
Fatigue assessment | It is assessed at baseline and after 24 hours for each condition (capsaicin or placebo).
  Modified Fatigue Impact Scale (MFIS). The MFIS evaluates the degree to which fatigue influences overall perceived function over the last 4 weeks. It assesses three subscales: cognitive (9 items), physical (10 items), and psychosocial (2 items) functioning. Items are measured on a scale from 0 = "no problem" to 4 = "extreme problem", with a maximum score of 120. Higher scores indicate higher levels of fatigue.
Positive and negative affect | They are assessed at baseline and after 24 hours for each condition (capsaicin or placebo).
  Positive and Negative Affect Scale (PANAS). This scale consists of 20 items assessing two groups of emotions: negative and positive (10 items each). Subjects rate the intensity of a specific emotion they are experiencing at the moment on a scale (1 = "very slightly or not at all" to 5 = "Extremely"). for each emotion group with a maximum of 50. Higher scores indicate more intense emotions. The positive affect items were "interested," "excited," "strong," "enthusiastic," "proud," "alert," "inspired," "determined," "attentive," and "active." The negative affect items were "distressed," "upset," "guilty," "scared," "hostile," "irritable," "ashamed," "nervous," "jittery," and "afraid."
Depression scores | They are assessed at baseline and after 24 hours for each condition (capsaicin or placebo).
  Beck Depression Inventory (BDI-II). The BDI determines the severity of depressive mood states and consists of 21 questions assessing hopelessness, guilt, fatigue, and other physical symptoms, rated between 0 = "no symptom impact" and 3 = "maximum symptom impact" with a maximum score of 63. Higher scores indicate severe depressive symptoms. To obtain measures of trait depression, subjects in this study are instructed to rate the items in relation to how they generally feel.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Graven-Nielsen, DMSc, PhD, Study Director — Aalborg University
Locations (1):
- Aalborg University, Department of Health Sciences and technology, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
No personal data will be shared